CLINICAL TRIAL: NCT03426592
Title: Effect of High Dose Vitamin D Supplementation on HIV Latency: A Pilot Randomized Controlled Trial
Brief Title: Effect of High Dose Vitamin D Supplementation on HIV Latency
Acronym: VIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Melbourne Health (Other); The Alfred (Other); Melbourne Sexual Health Centre (Unknown); University of Illinois at Chicago (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Sharon Lewin, Director, The Peter Doherty Institute for Infection and Immunity, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016.362
Record Dates: First submitted 2018-02-01; First posted 2018-02-08 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Inflammation; Vitamin D; Immunomodulation; Virus latency
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Inflammation | interventions — Cholecalciferol; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3, 10000 Intl Units Oral Capsule (Active Comparator): Vitamin D3, 10000 Intl Units Oral Capsule, daily for 6 months
  Interventions: Drug: Vitamin D3, 10000 Intl Units Oral Capsule
- Placebo oral capsule (Placebo Comparator): Oleic acid capsule by mouth, daily for 6 months
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Vitamin D3, 10000 Intl Units Oral Capsule — Vitamin D capsule. Over-encapsulated to mimic placebo oral capsule.
  Eligible study participants will be randomized 1:1 to vitamin D or placebo one capsule daily from week 0 to week 24. All participants will be advised to achieve 1 gram daily dietary calcium intake whilst on study.
  Blood and urine will be taken at 0, 12, 24 and 36 weeks to evaluate the primary and secondary endpoints.
  Rectal swabs will be taken at 0, 24 and 36 weeks.
  All participants will continue antiretroviral therapy throughout the study.
  Other Names: Treatment Group
  Arms: Vitamin D3, 10000 Intl Units Oral Capsule
Drug: Placebo oral capsule — Capsule containing oleic acid. Over-encapsulated to mimic vitamin D3 capsule.
  Eligible study participants will be randomized 1:1 to vitamin D or placebo one capsule daily from week 0 to week 24. All participants will be advised to achieve 1 gram daily dietary calcium intake whilst on study.
  Blood and urine will be taken at 0, 12, 24 and 36 weeks to evaluate the primary and secondary endpoints.
  Rectal swabs will be taken at 0, 24 and 36 weeks.
  All participants will continue antiretroviral therapy throughout the study.
  Other Names: Control Group
  Arms: Placebo oral capsule

SUMMARY:
HIV persists despite antiretroviral therapy (ART) and is associated with chronic inflammation. This inflammation is thought to prevent an effective immune response against the virus and is mediated at least in part by gut epithelial permeability and microbial translocation. HIV accumulates preferentially within Th17 cells with time on ART; these memory CD4+ T cells are highly susceptible to HIV infection and are concentrated within the gut. Vitamin D promotes gut epithelial integrity in animal models and exerts anti-inflammatory effects on the human immune system including down-modulation of Th17 cell frequency. This study will evaluate whether high dose vitamin D is able to reduce immune activation and Th17 cell frequency, to improve gut barrier integrity and the gut microbiome and reduce HIV persistence in participants on long-term suppressive ART.

DETAILED DESCRIPTION:
The major barrier to a cure for HIV infection is the persistence of latently infected CD4+ T cells on antiretroviral therapy (ART). HIV is concentrated in vivo in Th17 cells in blood and the gastrointestinal tract. Th17 cells are critical mediators of mucosal immunity against bacteria and fungi and are rapidly depleted in the gut following HIV acquisition with subsequent gut epithelial permeability, microbial translocation and ensuing chronic inflammation which is not completely reversed on ART. Such inflammation may contribute to HIV persistence by potentiating T cell proliferation and thereby clonal expansion of infected cells, by exacerbating CD8+ T cell exhaustion and potentially by promoting viral replication despite ART.

Vitamin D has pleiotropic effects on the immune system including directing naïve CD4+ T cells away from the Th17 phenotype toward an anti-inflammatory regulatory T cell phenotype. It may also have beneficial effects on dendritic cell and CD8+ T cell immunity. Furthermore, vitamin D has been shown in animal models to strengthen gut epithelial integrity and in healthy volunteers to promote a more diverse gut microbiome.

The investigators plan to perform a pilot randomized double-blind placebo-controlled trial of high dose vitamin D supplementation in HIV-infected participants on suppressive ART and to determine its effect on immune activation, Th17 cell frequency, gut barrier integrity, the gut microbiome and HIV persistence.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* At least 18 years of age
* Documented HIV-1 infection
* Receiving combination antiretroviral therapy continuously for at least 3 years
* Viral load suppressed below 40 copies/mL, or below assay limit of quantification where limit of quantification is above 40 copies/mL, for at least 3 years (excluding single episodes of HIV viral load 40-500 copies/mL where subsequent viral load was below 40 copies/mL or below assay limit of quantification where limit of quantification is above 40 copies/mL)
* Viral load < 40 copies/ml at screening
* Screening 25-hydroxyvitamin D level within 12 months prior to recruitment between 50nM and 125nM
* Agreement not to take any vitamin D containing compounds other than study drug between screening and conclusion of the study
* Agreement not to have vitamin D level checked by a treating doctor during the study unless medically required

Exclusion Criteria:

* Any planned change to ART regimen within next 12 months (other than switching tenofovir disoproxil fumarate to tenofovir alafenamide)
* Known current acute or chronic hepatitis B, known current acute or chronic hepatitis C or positive HBsAg or HCV PCR in blood at screening
* Completion of curative treatment for HCV within 6 months prior to screening
* HIV-2 infection
* Any vitamin D supplementation from 6 months prior to the screening 25(OH) vitamin D test until study commencement (including multivitamins containing vitamin D and cod liver oil)
* Any medical indication for vitamin D supplementation, eg osteoporosis, renal impairment (estimated glomerular filtration rate < 60ml/minute), liver cirrhosis
* Chronic diarrhoea or fat malabsorption
* Body mass index (BMI >= 35)
* Current hypercalcaemia (corrected calcium greater than 2.60mM), current primary hyperparathyroidism or any history of nephrolithiasis
* Current hyperthyroidism
* History of sarcoidosis or active tuberculosis
* Grade 3 or 4 abnormalities in screening pathology laboratory tests not already excluded by the above criteria at the discretion of the Principal Investigator
* Hypersensitivity to vitamin D preparations
* Concurrent medication with adverse interactions with vitamin D (eg oral glucocorticoids, phenytoin, carbamazepine, barbiturates, rifampicin, rifabutin, St John's wort, thiazide diuretics, digoxin, ketoconazole, itraconazole, nefazodone, isoniazid, cholestyramine, aluminium hydroxide, aripiprazole, danazol, orlistat, perhexiline or sucralfate use) or possible such use within next 12 months
* Current interferon, immune checkpoint blocker, histone deacetylase inhibitor, oral vitamin A or other oral vitamin A analogue (eg acitretin, isotretinoin or tretinoin, also known as all-trans retinoic acid or ATRA) usage or possible use within next 12 months
* Current participation in another interventional HIV cure study
* Pregnancy or breast-feeding
* Participants of child-bearing potential unwilling to use at least one form of effective contraception (with failure rate <1%, eg hormonal contraception, intrauterine device, abstinence, tubal ligation or partner with vasectomy) from at least 2 weeks prior to study commencement until at least 4 weeks after discontinuation of all study medication
* Inability to consent
* Inability to speak English
* Medicare ineligibility
* Major medical or psychiatric illness or substance misuse that could in the opinion of the investigator impair adherence to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Change in total HIV DNA level | weeks 0 and 24
  The difference between the vitamin D and placebo arms in the mean change in frequency of total HIV DNA within CD4+ T cells from week 0 to week 24

SECONDARY OUTCOMES:
Change in other DNA markers of HIV persistence | Weeks 0, 12, 24, 36
  Total HIV DNA, integrated HIV DNA and 2-LTR circles in peripheral blood CD4+ T cells using PCR
Change in cell-associated HIV RNA | Weeks 0, 12, 24, 36
  Cell-associated unspliced and multiply spliced HIV RNA in peripheral blood CD4+ T cells using RT-PCR and Tat/rev Induced Limiting Dilution Assay (TILDA)
Change in proportion of immune cells | Weeks 0, 12, 24, 36
  T helper and T cytotoxic subsets, monocytes, dendritic cells and natural killer cells using flow cytometry
Change in T cell subset phenotype | Weeks 0, 12, 24, 36
  T cell subset activation and exhaustion marker and chemokine receptor expression using flow cytometry
Change in HIV-specific immunity | Weeks 0, 12, 24, 36
  HIV-specific CD4+ and CD8+ T cell frequency and polyfunctionality using HIV peptides and flow cytometry
Change in CD4+ T cell transcriptional profile | Weeks 0, 12, 24, 36
  CD4+ T cell transcriptional profile using RNA Seq
Change in high sensitivity C-reactive protein (hsCRP) | Weeks 0, 12, 24, 36
  hsCRP levels
Change in gut barrier permeability | Weeks 0, 12, 24, 36
  Gut barrier permeability using plasma lipopolysaccharide (LPS), soluble CD14 and intestinal fatty acid binding protein (I-FABP)
Change in gut microbiome diversity | Weeks 0, 24, 36
  Gut microbiome diversity using 16S rRNA sequencing and metagenomics
Change in plasma microbiome abundance and diversity | Weeks 0, 24, 36
  Plasma microbiome abundance and diversity using deep sequencing
25-hydroxyvitamin D levels | Weeks 0, 12, 24, 36
  Serum 25-hydroxyvitamin D levels and correlation between level achieved and each of the other endpoints (efficacy analysis)
Serum calcium levels | Weeks 0, 12, 24, 36
  Serum calcium corrected for albumin
Urinary calcium levels | Weeks 0, 12, 24, 36
  Urinary calcium:creatinine ratios and, where these are abnormal, 24 hour urinary calcium levels
Adverse events | Weeks 0, 12, 24, 36
  Incidence and severity of adverse events
Study protocol adherence | Weeks 0 to 24
  Adherence to study drug and 1g daily dietary calcium intake as measured by pill count and participant report

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lewin, FRACP PhD, Principal Investigator — The Peter Doherty Institute for Infection and Immunity, University of Melbourne
Locations (4):
- Australia (4):
  - The Peter Doherty Institute for Infection and Immunity, Melbourne, Victoria
  - The Alfred Hospital - Department of Infectious Diseases, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Melbourne Sexual Health Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pitman MC, Meagher N, Price DJ, Rhodes A, Chang JJ, Scher B, Allan B, Street A, McMahon JH, Rasmussen TA, Cameron PU, Hoy JF, Kent SJ, Lewin SR. Effect of high dose vitamin D3 on the HIV-1 reservoir: A pilot randomised controlled trial. J Virus Erad. 2023 Aug 29;9(3):100345. doi: 10.1016/j.jve.2023.100345. eCollection 2023 Sep. PMID 37753336